CLINICAL TRIAL: NCT04164485
Title: Clinical Study of Functional Collagen Scaffold Transplantation for Laryngeal Soft Tissue Regeneration
Brief Title: Functional Collagen Scaffold for Laryngeal Soft Tissue Regeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAS-XDA-LSTR/IGDB
Record Dates: First submitted 2019-10-31; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Glottic Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional collagen scaffold transplantation (Experimental)
  Interventions: Biological: Functional collagen scaffold transplantation
- Autologous adipose cell transplantation (Experimental)
  Interventions: Biological: Autologous adipose cell transplantation

INTERVENTIONS:
Biological: Functional collagen scaffold transplantation — Injectable collagen scaffold combined with autologous adipose-derived cells will be injected into submucosa of vocal cord and paraglottic space under the surgical microscope
  Arms: Functional collagen scaffold transplantation
Biological: Autologous adipose cell transplantation — Autologous adipose-derived cells will be injected into the submucosa of vocal cord and paraglottic space under the surgical microscope
  Arms: Autologous adipose cell transplantation

SUMMARY:
Unilateral vocal cord paralysis (UVCP) is a clinical condition and often leads to glottic insufficiency. The presence of glottic insufficiency can result in poor pronunciation quality, vocal fatigue, shortness of breath with speaking, and in some cases, it could lead to unable to pronounce, dysphagia and aspiration, severely decreasing quality of life for its victims. This study is carried out to explore the short-term and long-term efficacy of the functional collagen scaffold in guiding laryngeal soft tissue regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years old, male or female
2. Unilateral vocal cord injury and poor closure of the glottis
3. Disease course was more than 1 year
4. At least two GRBAS scores reach 2 points or more
5. The subjects have read and fully understood the research notes, signed informed consent

Exclusion Criteria:

1. Over speaking professionals, such as teachers, shop assistants
2. With vital organ dysfunction, such as heart, lung, liver or kidney
3. With malignant tumors
4. Pregnant or lactating women, or in preconception period
5. History of drug allergy
6. Difficult to be followed-up or cooperate long-termly
7. Participated in other clinical trials in the last 3 months
8. With severe progressive diseases
9. Alcoholics or drug addicts
10. Unable to execute clinical study protocol due to severe mental disorders or lingual barriers
11. With inevitable circumstances of voice damage
12. Any other unsuitable conditions for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
GRBAS scale | 1 week after intervention
  Auditory perceptual evaluation was assessed with a GRBAS scale, in which the voice properties, such as the grade of the severity of dysphonia (G), roughness (R), breathiness (B), asthenia (A), and strain (S), are scored on a four-point scale: 0 = normal, 1 = slight deviance, 2 = moderate deviance, and 3 = severe deviance
GRBAS scale | 1 month after intervention
  Auditory perceptual evaluation was assessed with a GRBAS scale, in which the voice properties, such as the grade of the severity of dysphonia (G), roughness (R), breathiness (B), asthenia (A), and strain (S), are scored on a four-point scale: 0 = normal, 1 = slight deviance, 2 = moderate deviance, and 3 = severe deviance
GRBAS scale | 3 month after intervention
  Auditory perceptual evaluation was assessed with a GRBAS scale, in which the voice properties, such as the grade of the severity of dysphonia (G), roughness (R), breathiness (B), asthenia (A), and strain (S), are scored on a four-point scale: 0 = normal, 1 = slight deviance, 2 = moderate deviance, and 3 = severe deviance
GRBAS scale | 6 month after intervention
  Auditory perceptual evaluation was assessed with a GRBAS scale, in which the voice properties, such as the grade of the severity of dysphonia (G), roughness (R), breathiness (B), asthenia (A), and strain (S), are scored on a four-point scale: 0 = normal, 1 = slight deviance, 2 = moderate deviance, and 3 = severe deviance
GRBAS scale | 9 month after intervention
  Auditory perceptual evaluation was assessed with a GRBAS scale, in which the voice properties, such as the grade of the severity of dysphonia (G), roughness (R), breathiness (B), asthenia (A), and strain (S), are scored on a four-point scale: 0 = normal, 1 = slight deviance, 2 = moderate deviance, and 3 = severe deviance
GRBAS scale | 12 month after intervention
  Auditory perceptual evaluation was assessed with a GRBAS scale, in which the voice properties, such as the grade of the severity of dysphonia (G), roughness (R), breathiness (B), asthenia (A), and strain (S), are scored on a four-point scale: 0 = normal, 1 = slight deviance, 2 = moderate deviance, and 3 = severe deviance

SECONDARY OUTCOMES:
Voice handicap index (VHI) scale | 1 week, 1, 3, 6, 9, 12 month after intervention
  The Voice Handicap Index (VHI) is a 30-item test divided into 3 subscales that measure the functional, physical and emotional features of the disability caused by voice impairment was used for patient self-assessment. The subscale scores ranged from 0 to 40, and the total ranged from 0 to 120, with a higher score indicating a greater degree of disability
Jitter | 1 week, 1, 3, 6, 9, 12 month after intervention
  Acoustic voice analysis parameter. Jitter is for short and middle term pitch perturbation analysis
Shimmer | 1 week, 1, 3, 6, 9, 12 month after intervention
  Acoustic voice analysis parameter. Shimmer is for short and middle term amplitude perturbation analysis
Normalized noise energy (NNE) | 1 week, 1, 3, 6, 9, 12 month after intervention
  Acoustic voice analysis parameter. Normalized Noise Energy (NNE) is automatically computed from the voice signals using an adaptive comb filtering method performed in the frequency domain
Maximum phonation time (MPT) | 1 week, 1, 3, 6, 9, 12 month after intervention
  Acoustic voice analysis parameter. Maximum phonation time (MPT) represents the maximum time that an individual can sustain the vowel /a/ at a comfortable pitch and loudness
Physical status of vocal cords | 1 week, 1, 3, 6, 9, 12, 24 month after intervention
  The morphology of vocal cords (thin or fat, smooth or rough, plump or atrophy), motor function of vocal cords (normal, limited or fixed) and glottic closure (yes or no) were observed by fiber laryngoscopy
Volume of vocal cords | Baseline, 1 year, 2 year after intervention
  The volume of vocal cords was evaluated by Computed tomography (CT)

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China